CLINICAL TRIAL: NCT07220382
Title: PREoperative Targeted OnabotulinumtoXina Injection for Abdominal Wall Reconstruction: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Preoperative BOTOX® Injection for Large Ventral Hernia Repair
Acronym: PRETOX
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Joseph and Florence Mandel Family Foundation (Unknown)
Responsible Party: Principal Investigator, Lucas Beffa, Assistant Professor of Surgery, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-824
Record Dates: First submitted 2025-10-17; First posted 2025-10-23 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hernia Abdominal Wall; Botox Injection; Hernia Incisional Ventral; Hernia Repair With Compartment Syndrome; Hernia Surgery; Hernia; Hernia Incisional
Keywords: BOTOX; Ventral Hernia; Abdominal Wall Reconstruction; OnabotulinumtoxinA; Preoperative BOTOX; Primary Fascial Closure; Fascial Bridging; Transversus Abdominis Release; Posterior Component Separation
MeSH Terms: conditions — Hernia, Abdominal; Hernia; Incisional Hernia; Hernia, Ventral | interventions — Botulinum Toxins, Type A; Sodium Chloride; Injections; Saline Solution; Fluoridation; Abdominoplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will be blinded to the intervention drug (botulinumtoxin vs placebo). Radiologist(s) performing the injection will be blinded to the intervention drug.
  Surgeon(s) performing the hernia repair will be blinded to the intervention drug.
  Only study personnel and pharmacists who are not participating in a patient's surgery will know the randomization group (intervention or placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OnabotulinumtoxinA Group (Experimental): These patients will receive image-guided botulinumtoxin injections as described 21-48 days prior to open ventral hernia repair.
  Interventions: Procedure: OnabotulinumtoxinA Injection; Drug: OnabotulinumtoxinA; Procedure: Open Ventral Hernia Repair
- Placebo Group (Placebo Comparator): These patients will receive image-guided saline (placebo) injections as described 21-48 days prior to open ventral hernia repair.
  Interventions: Procedure: Saline (placebo) Injection; Drug: 0.9 % Normal Saline; Procedure: Open Ventral Hernia Repair

INTERVENTIONS:
Procedure: OnabotulinumtoxinA Injection — A total of 300 units of onabotulinumtoxinA will be reconstituted 150 cc of injectable 0.9% NaCl (for a final concentration of 2 units / cc). Each side of the abdominal wall will receive a total 75 cc distributed across three injection sites (six injection sites total per patient). At each injection site, the muscle bodies of the transversus abdominis, internal oblique, and external oblique will receive an equivalent volume of product under ultrasonic or radiographic visualization.
  Other Names: BOTOX® Injection
  Arms: OnabotulinumtoxinA Group
Procedure: Saline (placebo) Injection — 150 cc of injectable 0.9% NaCl will be prepared. Each side of the abdominal wall will receive a total 75 cc distributed across three injection sites. At each injection site, the muscle bodies of the transversus abdominis, internal oblique, and external oblique will receive an equivalent volume of product under ultrasonic or radiographic visualization.
  Arms: Placebo Group
Drug: OnabotulinumtoxinA — 300 units of onabotulinumtoxinA will be prepared and administered as described in: "Procedure/Surgery: OnabotulinumtoxinA Injections"
  Other Names: BOTOX®
  Arms: OnabotulinumtoxinA Group
Drug: 0.9 % Normal Saline — 150cc of normal saline will be prepared and administered as described in: "Procedure/Surgery: Saline (placebo) Injection".
  Other Names: Saline; Salt Water; Placebo; Normal Saline; NaCl
  Arms: Placebo Group
Procedure: Open Ventral Hernia Repair — Open abdominal wall reconstruction will be conducted in our standard fashion for the repair of very large hernias. The surgery is the same for patients who are not in the study. Surgeons will be blinded to the study arm of participant patients.
  Other Names: Abdominal Wall Reconstruction; Posterior Component Separation

SUMMARY:
This study is for adults who need open surgery to repair a very large abdominal (ventral) hernia. This study tests whether a one-time, image-guided injection of a medicine commonly known as "BOTOX®" (onabotulinumtoxinA) into the side abdominal muscles 3-7 weeks before surgery helps surgeons close the abdominal wall fully at the end of the operation. Closing the muscle and tissue layers ("primary fascial closure") is linked to fewer problems after surgery and better quality of life.

Participants will be randomly assigned (like a coin flip) to receive either the BOTOX® medicine or a saltwater (placebo) injection. Neither patients nor the care team will know which one was given. All participants will still have their planned hernia repair in the standard way that we repair patients who are not part of the study. The study will track whether the abdomen can be closed without leaving a gap, and investigators will also look at recovery, complications, time in the ICU or on a ventilator, length of stay, pain, and quality-of-life scores. Most information will be collected during participants' hospital stay, but the investigators will continue to see how participants are doing up to 2 years after surgery. Short phone check-ins will occur before surgery, and after surgery follow-up happens around 30 days, 90 days, 1 year, and 2 years.

Possible risks from the injection include temporary muscle weakness, trouble swallowing or breathing, pain or infection at the injection site, and (if CT is used for guidance) a small amount of radiation exposure. Surgery itself carries the usual risks (pain, bleeding, wound problems). Benefits are not guaranteed, but the injection may make closure easier and recovery smoother. About 188 people will take part at Cleveland Clinic.

DETAILED DESCRIPTION:
Background and Rationale:

Massive ventral hernias (pre-op axial width ≥15 cm and/or Tanaka volume ratio >25%) seldom achieve primary fascial closure (PFC) and are associated with higher respiratory morbidity, intensive care unit (ICU) utilization, post-operative pain, hospital length of stay (LOS), cost, and recurrence. Spasticity/fibrosis of the external oblique-internal oblique-transversus abdominis (EO/IO/TA) complex likely limits lateral abdominal wall compliance and impedes midline medialization. Pre-operative, image-guided onabotulinumtoxinA (BOTOX®) has been proposed to elongate the lateral wall, enlarge the functional abdominal domain, reduce closure pressures, and thereby increase the primary fascial closure (PFC) rate. Prior institutional data show ~77% PFC in this population without pre-op toxin, whereas retrospective series suggest ~95% with toxin utilization, motivating a definitive randomized trial.

Design:

Single-center, randomized, double-blind, placebo-controlled superiority trial. Randomization uses pre-generated block allocation (statistician-generated). Analyses will be intention-to-treat (ITT), with a parallel per-protocol (PP) analyses limited to participants who receive the assigned injection and undergo AWR within 21-48 days post-injection. A single interim analysis is planned at 50% completion of primary endpoint. Intention-to-treat (ITT) is primary method of analysis; however, a per-protocol (PP) analysis will also be conducted as this supports causal inference among adherent participants. An independent DMC will review interim results and advise on continuation/early stopping.

Interventions:

Fully described in 'Arms and Interventions' section. Participants will either receive image-guided injections of BOTOX® at six sites on the lateral abdominal wall (three sites per side) with a total of 300 units give (2 u / cc concentration; 25 cc at each site); or, participants will receive the same volume of a 0.9% saline solution (25 cc at each site).

End Points and Outcomes:

Fully described in the 'Outcomes Measures' section. Primary endpoint is primary fascial closure (PFC), the successful closure of hernia defect at the conclusion of the case. Additional secondary outcomes regarding clinical course and patient-reported outcomes will be captured at 30 days, 90 days, 1 year, and 2 years.

Exploratory outcomes include cost and healthcare utilization information, as well as comparison of physiological parameters between treatment groups.

Data Stewardship:

Primary data capture occurs in the ACHQC registry, supplemented by an institutional REDCap database for variables not routinely captured (e.g., physiologic measures) in the registry.

ELIGIBILITY:
Inclusion Criteria:

* Adult (greater than or equal to 18 years of age)
* Candidate for elective open repair of ventral hernia
* Preoperative imaging demonstrating either:
* ventral hernia defect width of at lest 15 cm; AND/OR,
* Tanaka volume ratio of at least 25%
* Planned elective hernia repair in an open fashion via a midline laparotomy with posterior component separation and transversus abdominis release

Exclusion Criteria:

* Emergent cases
* Pregnancy and/or breastfeeding at time of intramuscular injection
* Inability to provide informed consent
* Inability to receive either study intervention (i.e. allergy to local anesthetics utilized for intervention administration, allergy and/or contraindication to any botulinum toxin, inability to attend outpatient administration of study intervention, inability to conform to safety check schedule)
* Known congenital or acquired neuromuscular disorder
* Presence of stoma
* Current infection at time of intramuscular injection
* Flank hernias s defined by EHS L1-L4
* BMI > 45 kg/m^2
* Diaphragmatic hemiparesis or chronic obstructive pulmonary disease (COPD) with chronic oxygen dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
Primary Fascial Closure (PFC) at conclusion of Hernia Surgery (Yes / No, determined by surgeon) | This will be measured (recorded) on the day of the hernia repair surgery, which will be 21 to 48 days after receiving your BOTOX injection.
  Primary fascial closure (PFC) is the successful closure of the hernia. It will be defined in a binary, categorical manner as: "Yes" (fascial closed) or "No" (fascia not closed and bridging mesh required). To be considered "Yes" for PFC, the midline anterior fascia must be completely re-approximated via absorbable running or figure-of-eight sutures. If any segment of the anterior fascia cannot be approximated and closed, the patient will require anterior bridging and this would be considered a failure of PFC.
  Surgeons will decide if the fascia can be closed or if it cannot be closed by their expertise and discretion. No prespecified criteria have been established which dictate operative decision-making. The study team will record an outcome of "Yes" for PFC if the fascia is successfully closed by the surgeon via an eligible technique as previously described.

SECONDARY OUTCOMES:
30-Day Surgical Site Occurrence (SSO) - Proportion of Participants (%) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  SSOs will be abstracted from the clinical record in a prospective fashion. They are defined as wound-related problems at or near the incision within 30 days of surgery (e.g., infection, fluid or blood collections, wound separation, or skin edge death). These will be measured on an individual level basis, and will be captured via patient interview and chart review within the specified timeframe. Aggregate calculation for a population: numerator = participants with ≥1 SSO; denominator = all randomized participants who underwent surgery; unit = participants (%).
30-Day Surgical Site Infection (SSI) - Proportion of Participants (%) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  Any incisional or organ/space infection within 30 days, identified by treating teams. These will be measured on an individual level basis, and will be captured via patient interview, clinician-report, and/or chart review within the specified timeframe. Defined via any antibiotic and/or antimicrobial treatment of an infection at the surgical site. Positive culture or proof of pathogen not needed. Aggregate calculation for a population: numerator = participants with ≥1 SSO; denominator = all randomized participants who underwent surgery; unit = participants (%).
30-Day SSOPI (Surgical Site Occurrence Requiring Procedural Intervention) - Proportion of Participants (%) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  These are SSO events (as described in 30-Day SSO outcome) that required a bedside/clinic or OR procedure (e.g., aspiration, drainage, debridement) within 30 days. Cumulative SSOPIs will be calculated for each group. Additionally, aggregate calculation for a study group: numerator = participants with ≥1 SSOPI; denominator = all randomized participants who underwent surgery; unit = participants (%).
30-Day Readmission - Proportion of Participants (%) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  Any inpatient hospital readmission within 30 days of index surgery. "How measured": EHR review/REDCap; unit = participants (%).
30-Day Reoperation - Proportion of Participants (%) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  Any return to the operating room related to the index surgery within 30 days. "How measured": EHR/REDCap; unit = participants (%).
30-Day Hospital Length of Stay - Days | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  Days from operation to hospital discharge. "How measured": EHR discharge date minus surgery date; unit = days.
30-Day ICU Admission - Proportion of Participants (%) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  Any ICU care during the index stay or within 30 days (planned or unplanned). "How measured": EHR/REDCap; unit = participants (%).
Duration of Mechanical Ventilation (Index Hospitalization) - Hours | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  Total ventilator time during and after surgery until final extubation during the index stay. Will be sub-divided as during surgery and after surgery. "How measured": anesthesia/intensive care record; unit = hours (may also be displayed as days:hours)
30-Day Myocardial Infarction (MI) - Proportion of Participants (%) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  MI within 30 days per treating clinician diagnosis. "How measured": medical record review, patient interview, and/or clinical diagnosis. Unit = participants (%).
30-Day Pneumonia - Proportion of Participants (%) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  Clinically diagnosed pneumonia within 30 days. "How measured": patient interview, medical record review, or clinical diagnosis. Unit = participants (%).
30-Day Renal Failure/Acute Kidney Injury (AKI) - Proportion of Participants (%) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  Acute kidney injury/failure within 30 days. "How measured": clinician diagnosis, medical record review, and/or KDIGO Guidelines. Unit = participants (%).
30-Day Post-operative Ileus - Proportion of Participants (%) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  Ileus requiring clinical management within 30 days. Defined as placement of an nasogastric tube or clinical diagnosis by surgeon based on intolerance of oral intake or delayed return of bowel function. "How measured": medical record review or clinician diagnosis. Unit = participants (%).
30-Day Patient-Reported Outcomes Measurement Information System (PROMIS®) Pain Intensity Short Form 3a - T-Score (Raw Response score range: 0-10, Higher = Worse Pain) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  Three-item pain intensity questionnaire. "How measured": PROMIS-3a administered at follow-up; raw sum (3-15) converted to T-score (mean 50, SD 10); higher scores = more pain (worse). Unit = T-score.
30-Day Hernia-Related Quality-of-Life Survey (HerQLes) - Score (0-100; Higher = Better QoL) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  12-item hernia-specific QoL instrument. "How measured": HerQLes administered at follow-up; score transformed 0-100, higher = better function/less disability. Unit = total score (0-100).
30-Day Complication Severity (Clavien-Dindo) - Distribution of Highest Grade (I-V) | Approximately 30 to 45 days after hernia repair surgery, which would be approximately 2 to 3 months after injection procedure.
  Highest complication grade based on the Clavien-Dindo classification system per participant within 30 days. "How measured": graded in REDCap from clinical documentation; unit = participants in each grade (%). Minimum = I, maximum = V; higher grades = worse.
90-Day SSO - Proportion of Participants (%) | Approximately 3 months after hernia repair surgery, which would be about 4 to 5 months after injection procedure.
  SSOs will be abstracted from the clinical record in a prospective fashion. They are defined as wound-related problems at or near the incision within 90 days of surgery (e.g., infection, fluid or blood collections, wound separation, or skin edge death). These will be measured on an individual level basis, and will be captured via patient interview and chart review within the specified timeframe. Aggregate calculation for a population: numerator = participants with ≥1 SSO; denominator = all randomized participants who underwent surgery; unit = participants (%).
90-Day SSI - Proportion of Participants (%) | Approximately 3 months after hernia repair surgery, which would be about 4 to 5 months after injection procedure.
  Any incisional or organ/space infection within 90 days, identified by treating teams. These will be measured on an individual level basis, and will be captured via patient interview, clinician-report, and/or chart review within the specified timeframe. Defined via any antibiotic and/or antimicrobial treatment of an infection at the surgical site. Positive culture or proof of pathogen not needed. Aggregate calculation for a population: numerator = participants with ≥1 SSO; denominator = all randomized participants who underwent surgery; unit = participants (%).
90-Day SSOPI - Proportion of Participants (%) | Approximately 3 months after hernia repair surgery, which would be about 4 to 5 months after injection procedure.
  These are SSO events (as described in 30-Day SSO outcome) that required a bedside/clinic or OR procedure (e.g., aspiration, drainage, debridement) within 90 days. Cumulative SSOPIs will be calculated for each group. Additionally, aggregate calculation for a study group: numerator = participants with ≥1 SSOPI; denominator = all randomized participants who underwent surgery; unit = participants (%).
90-Day Complication Severity (Clavien-Dindo) - Distribution of Highest Grade (I-V) | Approximately 3 months after hernia repair surgery, which would be about 4 to 5 months after injection procedure.
  Highest complication grade based on the Clavien-Dindo classification system per participant within 90 days. "How measured": graded in REDCap from clinical documentation; unit = participants in each grade (%). Minimum = I, maximum = V; higher grades = worse.
90-Day Comprehensive Complication Index (CCI) Score at 90 Days - Score | Approximately 3 months after hernia repair surgery, which would be about 4 to 5 months after injection procedure.
  Comprehensive Complication Index® score, which is a weighted score based on the number of complications in each Clavien-Dindo group within 90 postoperative days. "How measured": the individuals CCI score at 90-days, as calculated via https://www.cci-calculator.com/.
90-Day Readmission - Proportion of Participants (%) | Approximately 3 months after hernia repair surgery, which would be about 4 to 5 months after injection procedure.
  Any inpatient hospital readmission within 30 days of index surgery. "How measured": EHR review/REDCap; unit = participants (%).
90-Day Reoperation - Proportion of Participants (%) | Approximately 3 months after hernia repair surgery, which would be about 4 to 5 months after injection procedure.
  Any return to the operating room related to the index surgery within 90 days. "How measured": patient interview, medical record review, surgeon report; unit = participants (%).
90-Day Patient-Reported Outcomes Measurement Information System (PROMIS®) Pain Intensity Short Form 3a - T-Score (Raw Response score range: 0-10, Higher = Worse Pain) | Approximately 3 months after hernia repair surgery, which would be about 4 to 5 months after injection procedure.
  Three-item pain intensity questionnaire. "How measured": PROMIS-3a administered at follow-up; raw sum (3-15) converted to T-score (mean 50, SD 10); higher scores = more pain (worse). Unit = T-score.
90-Day Hernia-Related Quality-of-Life Survey (HerQLes) - Score (0-100; Higher = Better QoL) | Approximately 3 months after hernia repair surgery, which would be about 4 to 5 months after injection procedure.
  12-item hernia-specific QoL instrument. "How measured": HerQLes administered at follow-up; score transformed 0-100, higher = better function/less disability. Unit = total score (0-100).
1-Year Surgical Site Occurrence (SSO) - Proportion of Participants (%) | Approximately 1 year after hernia repair surgery
  SSOs will be abstracted from the clinical record in a prospective fashion. They are defined as wound-related problems at or near the incision within 1 year of surgery (e.g., infection, fluid or blood collections, wound separation, or skin edge death). These will be measured on an individual level basis, and will be captured via patient interview and chart review within the specified timeframe. Aggregate calculation for a population: numerator = participants with ≥1 SSO; denominator = all randomized participants who underwent surgery; unit = participants (%).
1-Year Surgical Site Infection (SSI) - Proportion of Participants (%) | Approximately 1 year after hernia repair surgery
  Any incisional or organ/space infection within 1 year, identified by treating teams. These will be measured on an individual level basis, and will be captured via patient interview, clinician-report, and/or chart review within the specified timeframe. Defined via any antibiotic and/or antimicrobial treatment of an infection at the surgical site. Positive culture or proof of pathogen not needed. Aggregate calculation for a population: numerator = participants with ≥1 SSO; denominator = all randomized participants who underwent surgery; unit = participants (%).
1-Year SSOPI - Proportion of Participants (%) | Approximately 1 year after hernia repair surgery
  These are SSO events (as described in 30-Day SSO outcome) that required a bedside/clinic or OR procedure (e.g., aspiration, drainage, debridement) within 1 year. Cumulative SSOPIs will be calculated for each group. Additionally, aggregate calculation for a study group: numerator = participants with ≥1 SSOPI; denominator = all randomized participants who underwent surgery; unit = participants (%).
1-Year Reoperation | Approximately 1 year after hernia repair surgery
  Any return to the operating room related to the index surgery within 1 year. "How measured": patient interview, medical record review, surgeon report; unit = participants (%).
1-Year Reoperation for Hernia Recurrence | Approximately 1 year after hernia repair surgery
  Any return to the operating room related repair of a hernia within 7 cm of the hernia repaired in the original surgery within 1 year. "How measured": patient interview, medical record review, surgeon report; unit = participants (%).
1-Year Hernia Recurrence (Clinical) | Approximately 1 year after hernia repair surgery
  A recurrence after hernia repair is defined as a new hernia detected within 7cm of the original repair. The hernia must be determined via imaging (ultrasound, computed tomography scan, or magnetic resonance imaging scan) or the documented physical exam of a licensed practitioner. Determined as within 1 year of the hernia repair surgery.
1-Year Hernia Recurrence (Patient-Reported) | Approximately 1 year after hernia repair surgery
  Patient self-reported concern for recurrence based on response to the the question, "Do you feel or see a bulge?" on the Ventral Hernia Recurrence Inventory (VHRI) questionnaire. Asked at 1 year.
1-Year Patient-Reported Outcomes Measurement Information System (PROMIS®) Pain Intensity Short Form 3a - T-Score (Raw Response score range: 0-10, Higher = Worse Pain) | Approximately 1 year after hernia repair surgery
  Three-item pain intensity questionnaire. "How measured": PROMIS-3a administered at follow-up; raw sum (3-15) converted to T-score (mean 50, SD 10); higher scores = more pain (worse). Unit = T-score.
1-Year Hernia-Related Quality-of-Life Survey (HerQLes) - Score (0-100; Higher = Better QoL) | Approximately 1 year after hernia repair surgery
  12-item hernia-specific QoL instrument. "How measured": HerQLes administered at follow-up; score transformed 0-100, higher = better function/less disability. Unit = total score (0-100).
2-Year Surgical Site Occurrence (SSO) - Proportion of Participants (%) | Approximately 2 years after hernia repair surgery
  SSOs will be abstracted from the clinical record in a prospective fashion. They are defined as wound-related problems at or near the incision within 2 years of surgery (e.g., infection, fluid or blood collections, wound separation, or skin edge death). These will be measured on an individual level basis, and will be captured via patient interview and chart review within the specified timeframe. Aggregate calculation for a population: numerator = participants with ≥1 SSO; denominator = all randomized participants who underwent surgery; unit = participants (%).
2-Year Surgical Site Infection (SSI) - Proportion of Participants (%) | Approximately 2 years after hernia repair surgery
  Any incisional or organ/space infection within 2 years, identified by treating teams. These will be measured on an individual level basis, and will be captured via patient interview, clinician-report, and/or chart review within the specified timeframe. Defined via any antibiotic and/or antimicrobial treatment of an infection at the surgical site. Positive culture or proof of pathogen not needed. Aggregate calculation for a population: numerator = participants with ≥1 SSO; denominator = all randomized participants who underwent surgery; unit = participants (%).
2-Year SSOPI - Proportion of Participants (%) | Approximately 2 years after hernia repair surgery
  These are SSO events (as described in 30-Day SSO outcome) that required a bedside/clinic or OR procedure (e.g., aspiration, drainage, debridement) within 2 years. Cumulative SSOPIs will be calculated for each group. Additionally, aggregate calculation for a study group: numerator = participants with ≥1 SSOPI; denominator = all randomized participants who underwent surgery; unit = participants (%).
2-Year Reoperation | Approximately 2 years after hernia repair surgery
  Any return to the operating room related to the index surgery within 2 years. "How measured": patient interview, medical record review, surgeon report; unit = participants (%).
2-Year Reoperation for Hernia Recurrence | Approximately 2 years after hernia repair surgery
  Any return to the operating room related repair of a hernia within 7 cm of the hernia repaired in the original surgery within 2 years. "How measured": patient interview, medical record review, surgeon report; unit = participants (%).
2-Year Hernia Recurrence (Clinical) | Approximately 2 years after hernia repair surgery
  A recurrence after hernia repair is defined as a new hernia detected within 7cm of the original repair. The hernia must be determined via imaging (ultrasound, computed tomography scan, or magnetic resonance imaging scan) or the documented physical exam of a licensed practitioner. Determined as within 2 years of the hernia repair surgery.
2-Year Hernia Recurrence (Patient-Reported) | Approximately 2 years after hernia repair surgery
  Patient self-reported concern for recurrence based on response to the the question, "Do you feel or see a bulge?" on the Ventral Hernia Recurrence Inventory (VHRI) questionnaire. Asked at 2 years.
2-Year Patient-Reported Outcomes Measurement Information System (PROMIS®) Pain Intensity Short Form 3a - T-Score (Raw Response score range: 0-10, Higher = Worse Pain) | Approximately 2 year after hernia repair surgery
  Three-item pain intensity questionnaire. "How measured": PROMIS-3a administered at follow-up; raw sum (3-15) converted to T-score (mean 50, SD 10); higher scores = more pain (worse). Unit = T-score.
2-Year Hernia-Related Quality-of-Life Survey (HerQLes) - Score (0-100; Higher = Better QoL) | Approximately 2 year after hernia repair surgery
  12-item hernia-specific QoL instrument. "How measured": HerQLes administered at follow-up; score transformed 0-100, higher = better function/less disability. Unit = total score (0-100).

OTHER OUTCOMES:
Fascial Tension (Pre-Release and Post-Component Separation) - Force Units (lbs) | During hernia repair surgery
  Force required to bring each fascial edge to midline, measured twice: (1) after initial dissection/before retro-rectus release and (2) after each step during posterior component separation. "How measured": sterile Kocher clamps attached to fascia will be connected to a sterilizable tensiometers which is pulled until midline is reached by medial fascial edge; force recorded. Unit = pounds of force (lbs); higher values = greater tension.
Plateau Airway Pressure - cmH₂O | During hernia repair surgery and one day after surgery (if still requiring mechanical ventilation post-operatively)
  Ventilator plateau pressure measured (a) after intubation before incision, (b) just before skin closure (after repair), and (c) POD1 if still intubated. "How measured": volume-controlled ventilation; inspiratory pause 0.5-3 s; stabilized pressure recorded as Pplat; also record PIP, tidal volume, ventilator mode, PEEP, FiO₂. Unit = cmH₂O.
Change in Plateau Pressure With Closure - cmH₂O | During hernia repair surgery
  Difference between pre-closure and post-closure plateau pressures; negative change indicates improved mechanics. "How measured": subtraction of time-point values. Unit = cmH₂O.
Bladder Pressure (Intra-abdominal Pressure Proxy) - mmHg | During hernia repair surgery and one day after surgery (if foley remains in place)
  Measured three times for all patients: (1) after anesthesia before incision and (2) immediately pre-extubation; also (3) on POD1 prior to Foley removal. "How measured": per WSACS consensus - instill ≤25 mL sterile saline via stopcock into a clamped Foley; patient supine with bed flat; transduce at mid-axillary line at end-expiration. Unit = mmHg.
Abdominal Perfusion Pressure (APP) - mmHg | During hernia repair surgery and one day after surgery (if foley remains in place)
  Calculated as mean arterial pressure (MAP) - intra-abdominal pressure (from bladder pressure). "How measured": MAP (non-invasive or invasive, properly zeroed will be collected during regular care) and bladder pressure (as described above); APP computed. Unit = mmHg
Hernia Defect Size After Dissection - Width and Length (cm) | During hernia repair surgery
  Maximum width and length of the hernia defect following dissection/component separation. "How measured": intra-operative ruler measurement; unit = centimeters.
Anterior Fascial Defect Size When Bridging Required - Width and Length (cm) | During hernia repair surgery
  If PFC not achieved, the residual anterior defect dimensions at closure. "How measured": intra-op ruler; unit = cm.
Posterior Sheath Defect Size if Not Closed - Width and Length (cm) | During hernia repair surgery
  If posterior sheath cannot be closed, record dimensions. "How measured": intra-op ruler; unit = cm. Note: posterior bridging does not equal PFC failure.
Reason for Failure to Achieve Primary Fascial Closure - Frequency by Category | During hernia repair surgery
  Surgeon-reported reason(s) categorized and tallied (e.g., excessive tension, loss of domain, patient instability). "How measured": operative note; unit = participants per category (%).
Not Extubated at Case Conclusion - Proportion of Participants (%) | Immediately after hernia repair surgery
  Participants still intubated at the end of the operation. "How measured": anesthesia record; unit = participants (%).
Immediate Post-operative ICU Admission - Proportion of Participants (%) | Immediately after hernia repair surgery
  Direct transfer to ICU from OR/PACU after surgery. "How measured": disposition orders; unit = participants (%).
Unplanned ICU Admission Post-operatively - Proportion of Participants (%) | Immediately after hernia repair surgery
  ICU transfer after initial non-ICU disposition. "How measured": bed movement logs/orders; unit = participants (%).
Total Direct Hospital Cost Through 90 Days - US Dollars (USD) | 3 months after hernia repair surgery, which would be about 4 to 5 months after injection procedure.
  All-cause direct costs during the surgical global period (90 days). "How measured": institutional cost accounting; unit = USD.
Days Between Injection and Surgery - Days | Immediately after hernia repair surgery
  Interval from image-guided injection to operative date. "How measured": scheduling records; unit = days. (Target window 21-48 days.)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas R Beffa, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Patients will not be consented for the sharing of individual participant data outside of the Cleveland Clinic.